CLINICAL TRIAL: NCT04697485
Title: Polydiuretic Therapy for Heart Failure With Preserved Ejection Fraction and Diabetes Mellitus: A Pilot Trial
Brief Title: Polydiuretic Therapy for Heart Failure With Preserved Ejection Fraction and Diabetes Mellitus
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment and funding challenges
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sadiya Khan, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00213243
Record Dates: First submitted 2020-12-07; First posted 2021-01-06 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: HF - Heart Failure; Diabetes Mellitus
Keywords: HFpEF
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus | interventions — Bumetanide; Eplerenone

STUDY DESIGN:
Intervention Model Description: This will be a proof-of-concept, non-randomized, pilot study of patients with HFpEF and diabetes mellitus to receiving polydiuretic therapy (bumetanide 0.5 mg + eplerenone 25 mg + dapaglifozin 5 mg) on top of background therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Low-Dose, Triple Polydiuretic Therapy (LDTPT) (Experimental): Polydiuretic therapy will consist of bumetanide 0.5 mg + eplerenone 25 mg + dapaglifozin 5 mg once daily for 4 weeks.
  Interventions: Drug: Bumetanide 0.5 mg, dapaglifozin 5 mg, eplerenone 25 mg

INTERVENTIONS:
Drug: Bumetanide 0.5 mg, dapaglifozin 5 mg, eplerenone 25 mg — Low-Dose, Triple Polydiuretic Therapy (LDTPT) Treatment consists of:
  * Loop diuretic (bumetanide 0.5 mg)
  * Mineralocorticoid receptor antagonist (eplerenone 25 mg)
  * Sodium-glucose co-transporter 2 inhibitor (SGLT2i): Farxiga® (dapagliflozin) 5 mg

SUMMARY:
This is a single-center, non-randomzied pilot study investigating a combination of targeted therapies as possible treatment for heart failure with preserved ejection fraction (HFpEF).

The study interviention is a Low-Dose, Triple Polydiuretic Therapy (LDTPT, or polydiuretic) including loop diuretic (bumetanide), mineralocorticoid receptor antagonist (eplerenone), and Sodium-glucose co-transporter 2 inhibitors (SGLT2i) therapy (dapaglifozin).

DETAILED DESCRIPTION:
Patients with HFpEF and diabetes mellitus will receive polydiuretic therapy consisting of bumetanide 0.5 mg + eplerenone 25 mg + dapaglifozin 5 mg on top of background therapy. These medicines are currently FDA approved and recommended by clinical practice guidelines for the treatment of HFpEF (bumetanide, eplerenone) and diabetes mellitus (dapaglifozin).

This study is designed to evaluate if combination pharmacotherapies with synergistic or additive diuretic properties can improve adherence, treatment efficacy, and effectiveness with fewer side effects

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years old)
2. English speaker
3. Established diagnosis of NYHA Class II or III heart failure with preserved ejection fraction, which has been present for at least 2 months

   a. NB: Patients in which additional pharmacological or device therapy is contemplated, or should be considered, must not be enrolled until therapy has been optimized and is stable for ≥1 month.
4. NT-proBNP >600 pg/ml (or if hospitalized for heart failure within the previous 12 months, NT-proBNP ≥400 pg/ml) at enrolment (Visit 1)

   a. If concomitant atrial fibrillation at Visit 1, NT-proBNP must be ≥900 pg/ml (irrespective of history of heart failure hospitalization)
5. Type 2 diabetes mellitus, regardless of background insulin use

Exclusion Criteria:

1. Known contraindication to bumetanide, eplerenone, or dapagliflozin.
2. Symptomatic hypotension or systolic BP <95 mmHg at 2 out of 3 measurements at visit 1.
3. Current acute decompensated HF or hospitalization due to decompensated HF <4 weeks prior to enrolment.
4. Myocardial infarction, unstable angina, stroke or transient ischemic attack (TIA) within 12 weeks prior to enrollment.
5. HF due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy or uncorrected primary valvular disease.
6. Type 1 diabetes mellitus
7. Symptomatic bradycardia or second or third-degree heart block without a pacemaker.
8. Evidence of secondary cause of hypertension e.g., renal artery stenosis; significant renal impairment (eGFR <50 ml/min/1.73 m2), raised serum potassium (above lab normal limit of 5.5 mEq/L).
9. Women who are pregnant, breast feeding or of childbearing potential and are not using and do not plan to continue using medically acceptable form of contraception throughout the study (pharmacological or barrier methods).
10. Concomitant illness, physical impairment or mental condition which in the opinion of the study team / primary care physician could interfere with the conduct of the study including outcome assessment.
11. Participation in a concurrent interventional medical investigation or pharmacologic clinical trial. Patients in observational, natural history or epidemiological studies not involving an intervention are eligible.
12. Participant's responsible primary care or other responsible physician believes it is not appropriate for participant to participate in the study.
13. Inability or unwillingness to provide written informed consent.
14. Involvement in the planning and/or conduct of the study.
15. Receiving current treatment with sulfonylureas.
16. Unable to complete study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in NT-proBNP | 4 weeks
  Change in NT-proBNP after 4 weeks of treatment

SECONDARY OUTCOMES:
Change in Systolic and Diastolic Blood pressure | 4 weeks
  Change in blood pressure after 4 weeks of treatment
Change in body weight | 4 weeks
  Change in weight after 4 weeks of treatment
Compliance | 4 weeks
  Overall compliance with polydiuretic as assessed by pill count

CONTACTS AND LOCATIONS:
Overall Officials: Sadiya Khan, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided